CLINICAL TRIAL: NCT00135122
Title: Medication Overuse Headache: A Randomised Double Blind Study of Prednisolone or Placebo in Withdrawal Therapy (Phase 3), and a Randomised 1 Year Follow up by Neurologist or General Physician After Successful Withdrawal Therapy
Brief Title: Prednisolone in the Treatment of Withdrawal Headache in Probable Medication Overuse Headache
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Svein Gunnar Gundersen, Sorlandet hospital HF
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 70203
Record Dates: First submitted 2005-08-24; First posted 2005-08-25 (Estimated); Last update posted 2008-09-12 (Estimated); Status verified 2008-09

CONDITIONS: Headache
Keywords: migraine; analgesics; tension type headache
MeSH Terms: conditions — Headache; Migraine Disorders; Tension-Type Headache | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2 (Placebo Comparator): Placebo in six days
  Interventions: Drug: prednisolone

INTERVENTIONS:
Drug: prednisolone — Prednisolone 60mg day 1 and 2 , 40mg day 3 and 4 , 20mg day 5 and 6
  Other Names: Prednison, prednisolon

SUMMARY:
The purpose of this study is to determine whether prednisolone is more effective than placebo in the first six days after initiation of medication withdrawal therapy for a medication overuse headache. Another purpose is to study whether patients followed by a neurologist 1 year after withdrawal do better than patients followed by a general practitioner.

DETAILED DESCRIPTION:
Data published BoeMG,Mygland A,Salvesen R; Neurology 2007 Jul 3;69(1):26-31

ELIGIBILITY:
Inclusion Criteria:

* Chronic daily headache and medication overuse fulfilling International Headache Society (IHS)-II criteria

Exclusion Criteria:

* Pregnancy
* Age under 18 and over 70 years
* Major mental disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2003-09; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint was a calculated mean headache (MH), based on number of days with headache and mean intensity of headache during the first six days after withdrawal. | 6 days

SECONDARY OUTCOMES:
number of days with zero or mild headache, days with moderate to strong headache, days without headache, Use of antiemetic drugs ,staying drug-free during the entire period. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Salvesen, Professor, Study Chair — University of Tromso
Locations (1):
- Sørlandet Sykehus HF, Kristiansand, Vest-Agder, Norway

REFERENCES:
- [Result] Boe MG, Mygland A, Salvesen R. Prednisolone does not reduce withdrawal headache: a randomized, double-blind study. Neurology. 2007 Jul 3;69(1):26-31. doi: 10.1212/01.wnl.0000263652.46222.e8. Epub 2007 May 2. PMID 17475943